CLINICAL TRIAL: NCT06453772
Title: Effect of Using a Mathematical Model Based on pre-and Post-surgical Hemoglobin Differences to Determine the Volume to Aspirate in Primary Body Liposuction.
Brief Title: How to Predict Post-Surgical Bleeding and Hemoglobin in Liposuction?
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: LIPOSUCTION-24
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Bleeding; Surgery
Keywords: bleeding; abdominoplasty; Liposuction; Hemoglobin
MeSH Terms: conditions — Hemorrhage | interventions — Lipectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing liposuction
  Interventions: Procedure: Liposuction

INTERVENTIONS:
Procedure: Liposuction — Primary or secondary liposuction is performed by the surgical staff. The study analyzed variables including weight, height, BMI, preoperative hemoglobin, and aspirated volume. Additionally, preoperative hemoglobin (Hb), hematocrit (Hto), platelets, prothrombin time (Tp), partial prothrombin time (TpT), and International Normalized Ratio (INR) were evaluated. Hb and Hto levels were reassessed 24 hours post-surgery to monitor changes.

SUMMARY:
To evaluate the effect of using a mathematical model developed through pre- and post-surgical hemoglobins to predict the volume to aspirate in patients undergoing primary body liposuction.

DETAILED DESCRIPTION:
Postoperative anemia is a significant risk associated with liposuction, yet the scientific literature lacks detailed data on blood loss relative to the volume of fat removed. To address this, the investigators aimed to develop a mathematical formula predicting the decrease in postoperative hemoglobin (Hb post) based on preoperative hemoglobin (Hb pre), Body Mass Index (BMI), and the volume of fat suctioned. An observational, analytical, non-experimental, prospective study was conducted on liposuction patients to validate this predictive formula. Statistical analysis using Spearman's test showed that the results were statistically significant (P < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Patients of indistinct gender, operated on at the Centro Médico Nacional de Occidente for primary liposuction.
* Age between 18 to 60 years old
* Liposuction technique used: Super wet or Tumescent.
* Surgical procedure on any area of the body
* Large volume liposuction (> 5 L)
* Use of regional anesthesia

Exclusion Criteria:

* Presence of any of the following comorbidities: Systemic Arterial Hypertension or Diabetes Mellitus type 2.
* Performance of 2 or more procedures
* Use of medications (NSAIDs and/or coadjuvants that modify coagulation times).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing the first-time liposuction procedure, operated in the Plastic and Reconstructive Surgery Service
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Bleeding Predicting Method | 12 months
  Mathematical model based on pre-and post-surgical hemoglobins to further predict estimated bleeding

CONTACTS AND LOCATIONS:
Locations (2):
- Mexico (2):
  - National Western Speciality Hospital, Mexican Social Security Institute, Guadalajara, Jalisco
  - Western Medical Center, Mexican Institute of Social Security, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: Undecided